CLINICAL TRIAL: NCT04939831
Title: A Multicenter Noninferior Randomized Controlled Study Comparing the Efficacy of Laparoscopic Versus Abdominal Radical Hysterectomy for Cervical Cancer(Stage IB3,IIA2)
Brief Title: Laparoscopic or Abdominal Radical Hysterectomy for Cervical Cancer(Stage IB3,IIA2)
Acronym: LAUNCH 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Collaborators: Children's Hospital of Fudan University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Zhongshan Hospital (Other); RenJi Hospital (Other); Taizhou Hospital, Affiliated Cancer Hospital of the University of Chinese Academy of Sciences (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUOBGY2021-05
Record Dates: First submitted 2021-06-09; First posted 2021-06-25 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Abdominal Radical Hysterectomy; Laparoscopic Radical Hysterectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): the group of LRH
  Interventions: Other: Total Laparoscopic or Robotic Radical Hysterectomy
- 2 (Active Comparator): the group of ARH
  Interventions: Other: Total Abdominal Radical Hysterectomy

INTERVENTIONS:
Other: Total Laparoscopic or Robotic Radical Hysterectomy — Radical hysterectomy with bilateral pelvic lymph node dissection is performed as standard type C RH by Q-M classification, including cardinal ligaments divided at pelvic sidewall and uterosacral ligaments divided at near the sacral origin and the upper 1/4 to 1/3 of the vagina.
  Arms: 1
Other: Total Abdominal Radical Hysterectomy — Radical hysterectomy with bilateral pelvic lymph node dissection is performed as standard type C RH by Q-M classification, including cardinal ligaments divided at pelvic sidewall and uterosacral ligaments divided at near the sacral origin and the upper 1/4 to 1/3 of the vagina.
  Arms: 2

SUMMARY:
The purpose of this study is to confirm whether there is a difference between laparoscopic radical hysterectomy (LRH) and abdominal radical hysterectomy (ARH) in patient survival for Cervical Cancer (Stage IB3, IIA2).

DETAILED DESCRIPTION:
The purpose of this study is to compare LRH (or robotic-assisted) and ARH in patients with cervical cancer (Stage IB3, IIA2), by a multicenter stratified randomized controlled study, mainly including the following aspects:

1. To compare the differences in PFS and OS between patients receiving LRH and ARH.
2. To investigate whether PFS and OS in LRH can be improved by more rigorous specification of surgical details (including tumor-free principles and standard surgical scopes).
3. To assess postoperative complications and quality of survival.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of squamous carcinoma of the cervix, adenocarcinoma, squamous adenocarcinoma (Stage IB3,IIA2).
2. Age ≥ 21 years and ≤ 70 years.
3. Surgery type B and C (refer to Q-M surgical staging)
4. Normal range of liver and kidney function and blood count (specific details below) Hemoglobin > 60g/L Platelets > 70*109/L Leukocytes > 3*109/L Creatinine < 50mg/dL Transaminase abnormal indicators ≤ 3 Maximum value of transaminases not exceeding 3 times the corresponding normal value.
5. No history of other malignancies.
6. Non-pregnancy.
7. Physical strength classification: Karnofsky score ≥ 60;
8. Subjects voluntarily joined the study, signed the informed consent form, were compliant and cooperated with the follow-up.
9. No psychiatric disorders and other serious immune system disorders (e.g. lupus erythematosus, myasthenia gravis, HIV infection, etc.) (Note: Maximum diameter measurement of cervical lesions is based on PET-CT, or CT, or MRI)

Exclusion Criteria:

1. Those who are contraindicated for various surgeries and cannot undergo surgery.
2. Patients who have received pelvic/abdominal radiotherapy irradiation or neoadjuvant chemotherapy for cervical cancer.
3. Patients with recurrent cervical cancer
4. Patients with CT, MRI or PET-CT suggesting suspicious metastasis of pelvic lymph nodes with maximum diameter >2cm after further improvement of preoperative examination.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1104 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
the rate of OS at 5 years | 5 years from surgery
  Compare between groups(Cox proportional hazards model will be used to estimate the hazard ratio and 95% CI for the effect of treatment on the 5-year OS rate.)

SECONDARY OUTCOMES:
the rate of PFS at 5 years | 5 years from surgery
  The curves of PFS at 5 years will be estimated using the Kaplan-Meier method. The logrank test will be used to test the above hypothesis, the 5-year PFS rate difference and its 95% confidence interval (CI) for the comparison between the two groups will be estimated.

OTHER OUTCOMES:
Analysis of continuous outcomes | 1 years from surgery
  Compare these between groups(The continuous outcomes include operative duration(min), anesthesia time(min), blood loss during operation(ml), postoperative pain score and postoperative hospital stay(day). The outcomes with normal distribution will be summarised using mean and standard deviation (SD), while the outcomes with non-normal distribution will be summarised using median and interquartile. The differences in the outcomes and 95% CIs will be analysed by generalised linear model (GLM) with treatment as fixed effect and with normal distribution and identity link function.)
Analysis of binary outcomes | 5 years from surgery
  Compare these between groups(The intraoperative complications, postoperative complications, one-month and one-year postoperative quality of life and sexual life will be treated as binary outcomes and will be summarised by number (%) of participants with the event. The differences in the outcomes and 95% CIs will be analysed by GLM with treatment as fixed effect and with binomial distribution and identity link function.)
Safety analysis | 5 years from surgery
  Adverse events (AEs) will be summarised using the number of AEs, the number (%) of participants with AEs by groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Jiang, PHD, Principal Investigator — The Obstetrics and Gynecology Hospital of Fudan University
Locations (1):
- The Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu X, Yu H, Bai Y, Hou Y, Lou W, Wang X, Zhu T, Zhang Y, Hu W, Xue X, Zhu Z, Xiang L, Li J, Fang X, Gao S, Feng H, Diao W, Zhang H, Du M, Yan W, Qiu L, Feng H, Zhu S, Du Y, Jiang H. A multicenter noninferior randomized controlled study comparing the efficacy of laparoscopic versus abdominal radical hysterectomy for cervical cancer (stage IB3 and IIA2): study protocol of the LAUNCH 3 trial. Trials. 2023 Aug 18;24(1):542. doi: 10.1186/s13063-023-07573-w. PMID 37592299

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT04939831/Prot_SAP_000.pdf